CLINICAL TRIAL: NCT04239378
Title: Clinical, Radiographic and Histomorphometric Comparison of Autogenous Demineralized Dentin Matrix Versus Bovine-Derived Xenograft for Socket Preservation: A Randomised Controlled Clinical Trial
Brief Title: Comparison of Autogenous Dentin Matrix Versus Bovine-Derived Xenograft for Socket Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, PROFESSOR, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_101639
Record Dates: First submitted 2019-12-27; First posted 2020-01-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Alveolar Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group -Autogenous dentin matrix and collagen membrane (Experimental): Test group - After atraumatic tooth extraction , socket will be augmented with autogenous dentin matrix and covered with collagen membrane and sutures are placed.
  Interventions: Procedure: socket preservation
- Control group-bovine derived xenograft and collagen membrane (Active Comparator): control group- After atraumatic tooth extraction, socket will be augmented with bovine derived xenograft and covered with collagen membrane and sutures are placed.
  Interventions: Procedure: socket preservation

INTERVENTIONS:
Procedure: socket preservation — Autogenous dentin matrix and collagen membrane(test group) Bovine derived xenograft and collagen membrane (control group)

SUMMARY:
The present study is a human, prospective, randomised controlled clinical trial will be conducted to explore and compare the clinical, radiographic and histomorphometric outcome of autogenous demineralised dentin(DDM) versus bovine derived xenograft(DBM) for socket preservation procedure.

DETAILED DESCRIPTION:
* After local anesthesia a full thickness flap will be minimally reflected buccally and lingually around the tooth not exceeding 3mm apical to the alveolar crest.
* Tooth extraction will be performed using atraumatic extraction methods using Periotome.
* After extraction, the socket will be thoroughly curetted, inspected and irrigated with sterile saline solution.
* The socket satisfying the inclusion and exclusion criteria will be randomly allocated to either test or control group.
* Intra surgical measurements will be recorded.
* Socket preservation will be performed with either Demineralized dentin matrix DDM(TEST) or bovine derived xenograft DBM (CONTROL). Bone graft will be extended to the height of intra proximal bone.
* Collagen membrane will be placed over the grafted site extending approximately 3mm apical to buccal and lingual crest.
* Flaps will be approximated with sutures.

ELIGIBILITY:
Inclusion Criteria:

* Teeth indicated for extraction and subsequent implant placement
* Age group of 18 to 55 years
* Single rooted tooth indicated for extraction due to endodontic failure, caries or Fracture
* Presence of >2 mm keratinized tissue to allow flap management
* Extraction site should have adjacent tooth on either side
* Systemically healthy patients
* Class II or III extraction socket defects according to Hammerele and Jung(2008)
* Full mouth plaque score(FMPS)<25% at baseline.(PI)
* Full mouth bleeding score(FMBS)<25% at baseline. (BI)

Exclusion Criteria:

* .Presence of dehiscence or fenestration in any of the socket, more than 50% of bone loss in any of the socket walls
* Medical conditions contraindicating surgical interventions
* Known smokers and alcoholics
* Subjects with known bone metabolic disorders.(Pagets disease,fibrous dysplasia etc.)
* Acute infections at the site of extraction. Eg , Abscess
* History of malignancy
* Patients who have undergone radiotherapy or chemotherapy
* Periapical pathology such as granulomas, cyst, hypercementosis, ankylosis.
* Pregnant and lactating women
* Maxillary and mandibular 3rd molars.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Height of Alveolar Crest and Bucco-Lingual Ridge Width | 6 Months
  Using Mapping Caliper and (University of North Carolina) UNC- 15 PROBE Measured in mm
Alveolar Ridge Width Gain(ARWG) and Vertical Bone Height Gain(VBHG) | 6 MONTHS
  CBCT (Cone Beam Computer Tomography) measured in mm
New Bone Formation % and Residual Bone Graft | 6 MONTHS
  HISTOMORPHOMETRIC

SECONDARY OUTCOMES:
Plaque Index | 6months
  Silness and Leo index using UNC-15 PROBE with Rating Score Excellent- 0 Good- 0.1 - 0.9 Fair -1.0 - 1.9 Poor - 2.0 - 3.0
Bleeding Index | 6 months
  Mombelli - Sulcus Bleeding Index using UNC-15 Probe with Rating Score 0- No bleeding
  1 -Isolated bleeding spots visible 2-Blood forms a confluent red line on the margin 3- Heavy or profuse bleeding
Patient Reported Outcome Measures for Pain and Esthetics | 6 months
  ( Visual Analog Scale -VAS) Rating score, None (0) Mild (1-3) Moderate (4-6) Severe (7-10)

CONTACTS AND LOCATIONS:
Overall Officials: DR.JOANN PAULINE GEORGE, MDS, Principal Investigator — KRISHNADEVARAYA COLLEGE OF DENTAL SCIENCE
Locations (1):
- Krishnadevaray College of Dental Science and Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No